CLINICAL TRIAL: NCT06611969
Title: Effects of Inspiratory Muscle Training As a Complement to Usual Training on Respiratory Function and Performance in Amateur Athletes
Brief Title: Inspiratory Muscle Training in Amateur Athletes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Francisco Martínez Arnau, Associate Professor of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-FIS-3390079
Record Dates: First submitted 2024-09-13; First posted 2024-09-25 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Amateur Athletes
Keywords: inspiratory muscle training; respiratory function; performance; exercise
MeSH Terms: conditions — Respiratory Aspiration; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The evaluators are unaware of the assignment at all times. Outcomes assessor will discover group assigment after data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inspiratory muscle training (IMT) plus conventional training group (Experimental): IMT group will perform inspiratory muscle training in conjunction with the conventional marathon training plan
  Interventions: Procedure: Exercise
- Conventional training group (not-IMT) group (Active Comparator): The not-IMT group will follow only the conventional marathon training plan
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Exercise — The training programme will consist of 5 weekly sessions of aerobic work, strength and mobility, plus specific training of the inspiratory muscles, 3 times a week, at a load between 50 and 80% of the maximum inspiratory pressure of each participant, after re-education of their diaphragmatic ventilation.
  Arms: Inspiratory muscle training (IMT) plus conventional training group
Procedure: Exercise — The training programme will consist of 5 weekly sessions of aerobic work, strength and mobility.
  Arms: Conventional training group (not-IMT) group

SUMMARY:
The main objective of the study is to study the changes in FEV1 with the introduction of the specific inspiratory muscle training programme in the training programme of the popular athletes included. In addition, the secondary aims are to observe the differences in the respiratory capacities of the patients, in the vital signs, VO2 max, respiratory frequency and cardiac variability, as well as to assess the running performance of the participants.

Participants will be assigned to one of 2 study groups: IMT group (n=20) or not-IMT group (n=20) The IMT group will perform inspiratory muscle training in conjunction with the conventional marathon training plan. The not-IMT group will follow only the conventional marathon training plan. The study will be conducted over a 12 week period.

ELIGIBILITY:
Inclusion Criteria:

* Individuals willing to follow the 16-week running training plan
* Possibility of combining aerobic training with inspiratory muscle training
* Previous half marathon runner

Exclusion Criteria:

* - Exclusive or professional dedication to athletics
* Previous or current use of respiratory muscle training.
* Inadequate or health risk physical condition
* Significant chronic cardiorespiratory diagnoses (e.g. moderate-severe COPD).
* Neurological, muscular or neuromuscular problems that interfere with the ability to participate in tests and training protocols.
* Discontinuity in the performance of training.
* A terminal illness or any other major medical contraindication
* Lack of informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Expiratory forced volume in first second | Before starting the intervention and after its completion (12 weeks)
  FEV1, in liters/second, assessed by spirometry

SECONDARY OUTCOMES:
Hearth rate variability | From the beginning to the end of the programme, recorded on a daily basis.
  In miliseconds, assessed by hearth rate monitor
Hearth rate | From the beginning to the end of the programme, recorded on a daily basis.
  Maximal and specifically in rest, measured in beats per minute, assessed by heart rate monitor
Respiratory rate | From the beginning to the end of the programme, recorded on a daily basis.
  Measured in respirations per minute, estimated by the hearth rate monitor.
Running performance | From the beginning to the end of the programme, recorded on a daily basis.
  Measured by running pace (time per kilometre) and perceived exertion (modified Borg scale 0-10), recorded individually in a written register.
Maximal inspiratory pressure | Before starting the intervention and after its completion (12 weeks)
  MIP, in cmH2O, assessed by inspiratory manouever
Maximal consumption of oxygen | Before starting the intervention and after its completion (12 weeks)
  VO2 max, in ml/kg/min, estimated by heart rate monitor in training efforts.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Miguel Martínez Arnau, PhD, Study Director — Universitat de Valencia, Spain
Locations (1):
- Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No